CLINICAL TRIAL: NCT05416645
Title: Prevalence, Predictors, and Management of Gastroesophageal Reflux After Laparoscopic Sleeve Gastrectomy Multicentric Cohort Study
Brief Title: Prevalence, Predictors and Management of Gastroesophageal Reflux After Laparoscopic Sleeve Gastrectomy
Acronym: LSG-GERD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ayman El Nakeeb, clinical professor, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LSG
Record Dates: First submitted 2022-06-06; First posted 2022-06-13 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-01

CONDITIONS: Gastroesophageal Reflux
Keywords: laparoscopic sleeve gastrectomy; morbid obesity; GERD
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: Patients with morbid obesity who had LSG between January 2017 to January 2022were included in the trial, which was a multicenter cohort study.
Who Masked: Participant, Investigator
Masking Description: Patients with morbid obesity who had LSG between January 2017 to January 2022were included in the trial, which was a multicenter cohort study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients in group I (G1) had GERD (Active Comparator): Patients developed GERD after LSG
  Interventions: Procedure: patients with GERD after LSG
- Patients in group I (G2) had no GERD (Active Comparator): Patients not developed GERD after LSG
  Interventions: Procedure: patients with GERD after LSG

INTERVENTIONS:
Procedure: patients with GERD after LSG — patients with GERD after LSG
  Other Names: GERD after LSG

SUMMARY:
From January 2017 to January 2022, we looked at patients who had primary LSG and developed GERD. Before and after surgery, patients for LSG performed barium meal in Trendelenburg position and upper GIT endoscopy. Esophageal manometry and 24 h PH metery for patients who developed GERD.

DETAILED DESCRIPTION:
Patients with morbid obesity who had LSG between January 2017 to January 2022were included in the trial, which was a multicenter cohort study. Patients with morbid obesity, defined as a BMI of more than 40 or less than 35 with at least one comorbidity and ages ranging from 16 to 65, were patients' eligibility criteria for LSG. Patients under the age of 16 or over 65, as well as those with severe GERD, pregnancy, or inflammatory bowel disease, were excluded from the trial.

The data were recorded in a prospective manner in a computerized file, all patients signed the informed consent form after the description of the technique and possible postoperative morbidities.

Before and after surgery, patients for LSG performed barium meal in Trendelenburg position and upper GIT endoscopy. Esophageal manometry and 24 h PH metery for patients who developed GERD.

The study's purpose was to determine the prevalence of GERD symptoms, as well as potential predictors of GERD symptoms following LSG and how GERD symptoms were managed after LSG.

ELIGIBILITY:
Inclusion Criteria:

* Patients with morbid obesity defined as a BMI of more than 40 or
* BMI less than 35 with at least one comorbidity and
* ages ranging from 16 to 65, were patients'

Exclusion Criteria:

* Patients under the age of 16 or over 65,
* those with severe GERD,
* pregnancy, or
* inflammatory bowel disease,

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1537 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
GERD-Health-Related Quality of Life (GERD-HRQL) questionnaire | one month
  GERD-Health-Related Quality of Life (GERD-HRQL) questionnaire including GERD symptoms easch one scaled from 1 to 5 the less score the better out come (1 the best and 5 is the worset)

SECONDARY OUTCOMES:
Gastropexy | one month
  YES (WITH GASTROPEXY) OR NO (WITHOUT GASTROPEXY) .....RISK FACTORS AND PROTECTIVE FACTORS for GERD
smoking | one month
  YES (WITH SMOKING) OR NO (WITHOUT SMOKING)......RISK FACTORS AND PROTECTIVE FACTORS for GERD

CONTACTS AND LOCATIONS:
Overall Officials: Ayman El E Nakeeb, Principal Investigator — Mansoura University, Gastrointestinal Surgery Center
Locations (1):
- Ayman El Nakeeb, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the study protocol will be available for another researcher
Supporting Information: Study Protocol
Time Frame: available for any researcher at any time
Access Criteria: e-mail elnakeebayman@yahoo.com
URL: http://www.mans.edu.eg/

REFERENCES:
- [Result] Emile SH, Ghareeb W, Elfeki H, El Sorogy M, Fouad A, Elrefai M. Development and Validation of an Artificial Intelligence-Based Model to Predict Gastroesophageal Reflux Disease After Sleeve Gastrectomy. Obes Surg. 2022 Aug;32(8):2537-2547. doi: 10.1007/s11695-022-06112-x. Epub 2022 May 21. PMID 35596915
- [Result] Chue KM, Goh DWX, Chua CME, Toh BC, Ong LWL, Wong WK, Lim CH, Tan JTH, Yeung BPM. The Hill's Classification Is Useful to Predict the Development of Postoperative Gastroesophageal Reflux Disease and Erosive Esophagitis After Laparoscopic Sleeve Gastrectomy. J Gastrointest Surg. 2022 Jun;26(6):1162-1170. doi: 10.1007/s11605-022-05324-x. PMID 35445323
- [Result] Pavone G, Tartaglia N, Porfido A, Panzera P, Pacilli M, Ambrosi A. The new onset of GERD after sleeve gastrectomy: A systematic review. Ann Med Surg (Lond). 2022 Apr 5;77:103584. doi: 10.1016/j.amsu.2022.103584. eCollection 2022 May. PMID 35432994
- [Result] Sancho Moya C, Bruna Esteban M, Sempere Garcia-Arguelles J, Ferrer Barcelo L, Monzo Gallego A, Mirabet Saez B, Mulas Fernandez C, Albors Baga P, Vazquez Prado A, Oviedo Bravo M, Montalva Oron E. The Impact of Sleeve Gastrectomy on Gastroesophageal Reflux Disease in Patients with Morbid Obesity. Obes Surg. 2022 Mar;32(3):615-624. doi: 10.1007/s11695-021-05808-w. Epub 2022 Jan 20. PMID 35048247
- [Derived] El Nakeeb A, Aldossary H, Zaid A, El Sorogy M, Elrefai M, Attia M, Sewefy AM, Kayed T, Aldawsari MA, Al Dossari HM, Mohammed MM. Prevalence, Predictors, and Management of Gastroesophageal Reflux Disease After Laparoscopic Sleeve Gastrectomy: a Multicenter Cohort Study. Obes Surg. 2022 Nov;32(11):3541-3550. doi: 10.1007/s11695-022-06264-w. Epub 2022 Sep 10. PMID 36087223
- See also: mansoura university — http://www.mans.edu.eg/
- Available data/document: Study Protocol: post LSG GERD — http://www.mans.edu.eg/ — Postlaparoscopic sleeve gastrectomy